CLINICAL TRIAL: NCT00804245
Title: A Pilot Study of Use of 11C-Choline PET-CT in the Metastatic Evaluation of Patients With Newly Diagnosed High Risk Adenocarcinoma of the Prostate
Brief Title: C-11 Choline PET-CT Scan in Finding Metastases in Patients With Newly Diagnosed High-Risk Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00005483; P30CA012197 (NIH); CCCWFU-85207
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- radiolabeled choline tracer scans (Experimental): PET-CT scans supplemented with Choline 11 tracer
  Interventions: Procedure: needle biopsy; Drug: PET-CT scans supplemented with 11C-Choline tracer

INTERVENTIONS:
Procedure: needle biopsy — Biopsy of positive findings found on CT scan
Drug: PET-CT scans supplemented with 11C-Choline tracer — Use of 11C-Choline tracer to enhance diagnostic utility of 11C-Choline tracer

SUMMARY:
RATIONALE: New diagnostic procedures, such as C-11 choline PET-CT scan, may be effective in finding cancer that has spread to the bone and lymph nodes in patients with prostate cancer.

PURPOSE: This clinical trial is studying how well C-11 choline PET-CT scan works in finding metastases in patients with newly diagnosed high-risk prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the sensitivity and specificity of PET-CT scan using C-11 choline in detecting bone and lymph node metastases in patients with newly diagnosed high-risk adenocarcinoma of the prostate.

Secondary

* To perform semi-quantitative analysis of tracer uptake using standard uptake values and qualitative analysis using pure visual analysis.
* To develop an algorithm that includes the routine use of C-11 choline PET-CT scan for the staging of patients with prostate cancer at high risk of metastatic disease.
* To determine whether the presence of C-11 choline PET-CT scan positivity in these patients is predictive of outcomes, including biochemical relapse-free survival, time to development of clinically apparent metastases, time to local failure, and overall survival.
* To obtain tissue specimens from these patients for correlative studies and further evaluation.
* To obtain information regarding the feasibility and characteristics of C-11 choline PET-CT scan after androgen suppression.

OUTLINE: Patients undergo CT scan of the abdomen and pelvis with IV contrast and a bone scan. Patients also undergo a C-11 choline PET-CT scan*. In the case of any positive scan, patients undergo a needle biopsy. If the biopsy is negative for metastatic disease or if the biopsy is positive for metastatic disease in a draining lymph node region, patients receive radiotherapy and hormonal (antiandrogen) therapy. If the biopsy is positive for metastatic disease at any other site, patients receive hormonal therapy alone.

NOTE: *The first 10 patients enrolled on the study who have a positive PET-CT scan and positive biopsy undergo a second PET-CT scan at 6 months after the initial PET-CT scan.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Prior negative prostate biopsy allowed
* High-risk disease, as defined by one of the following:
* PSA ≥ 20 ng/mL
* Gleason score ≥ 8
* Digital rectal examination revealing ≥ T2c disease (tumor involving more than one half of one lobe of the prostate)
* Creatinine < 2.0 mg/dL
* Able to tolerate PET scan, CT scan, and bone scan
* Able to tolerate IV and oral contrast
* Willing to undergo biopsy of positive findings on PET-CT scan, CT scan, or bone scan

Exclusion Criteria:

* Other cancer within the past 5 years (except for nonmelanoma skin cancer)
* No prior radiotherapy, hormonal therapy, surgery (other than biopsy), or cryotherapy for prostate cancer Prior transurethral resection of the prostate allowed

Ages: 30 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2012-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Determination of utility of 11C-Choline in enhancing efficacy of Pet-CT scans | Approximately 1 year
  To determine the differential usefulness 11C-Choline during PET-CT to enhance diagnostic capability in evaluating metastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Garg, PhD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States